CLINICAL TRIAL: NCT00510133
Title: A Phase II Study of Active Immunotherapy With GRNVAC1, Autologous Mature Dendritic Cells Transfected With mRNA Encoding Human Telomerase Reverse Transcriptase, in Patients With Acute Myelogenous Leukemia in Complete Clinical Remission
Brief Title: A Study of Active Immunotherapy With GRNVAC1 in Patients With Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asterias Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRNVAC1 CP06-151
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GRNVAC1 (Experimental): Autologous dendritic cell vaccine
  Interventions: Biological: GRNVAC1

INTERVENTIONS:
Biological: GRNVAC1 — Autologous dendritic cell vaccine

SUMMARY:
This is a phase II study to evaluate the safety, feasibility and efficacy of immunotherapy with GRNVAC1 in patients with AML.

DETAILED DESCRIPTION:
This is a multicenter, open-label evaluation of feasibility, safety and immunotherapy in patients with AML in complete clinical remission. Patients will undergo leukapheresis prior to or shortly after completing consolidation chemotherapy. Dendritic cells will be transfected with the messenger RNA encoding human telomerase reverse transcriptase (hTERT) and a portion of the lysosome-associated membrane protein LAMP-1 (LAMP), matured, aliquoted, and cryopreserved. The final autologous vaccine product is referred to as GRNVAC1. Patients will be vaccinated with weekly for 6 weeks,will "rest" for 4 weeks, then will receive 6 boost injections, each administered every other week for 12 weeks. Patients will be followed every 4 weeks until Week 54, then every 3 months for 1 year, then every 6 months up to approximately 5 years from the first vaccination or until relapse/progression.

ELIGIBILITY:
Inclusion Criteria:

* AML in first complete remission (CR1) or in second complete remission (CR2) with CR1 >/= 6 months
* Has completed at least one cycle of consolidation chemotherapy within past 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hepatic/renal function

Exclusion Criteria:

* CR1 and good risk cytogenetic features [t(15;17), t(8;21), inv(16) or t(16:16)]
* Central nervous system or leptomeningeal disease
* Allogeneic stem cell transplant planned or expected
* Documented allergy to penicillin or beta-lactam antibiotics
* Active or ongoing autoimmune disease
* Clinically significant pulmonary or cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Feasibility will be assessed by examining whether enough cells are collected during leukapheresis, whether enough vaccine is manufactured for at least 2 injections, and whether the patient is still in remission when the vaccine is released. | 1 year

SECONDARY OUTCOMES:
Immunological response, defined as the proportion of patients with a positive induction of hTERT-specific T cells to twice the pre-vaccination level, the proportion of patients with DTH, and event-free survival. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John F DiPersio, MD,PhD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - Emory University School of Medicine, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ohio State University, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- See also: Related Info — http://www.geron.com